CLINICAL TRIAL: NCT04237428
Title: Clinical Study on the Treatment of Relapsed or Refractory CD19 Positive Non-Hodgkin's Lymphoma Patients With Target CD19 Chimeric Antigen Receptor T Cell Infusion
Brief Title: CD19-CART in the Treatment of R/R CD19 Positive Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-19-001
Record Dates: First submitted 2020-01-13; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hCD19 CAR-T cells Infusion (Experimental)
  Interventions: Biological: CD19 CAR-T cells infusion

INTERVENTIONS:
Biological: CD19 CAR-T cells infusion — Biological: CD19 CAR-T cells infusion Biological: CD19 CAR-T cells infusion. Pretreatment: patients enrolled in this study will receive cyclophosphamide or fludarabine plus cyclophosphamide. CD19 CAR-T cells infusion are allowed within 2 weeks after treatment.
  CD19 CAR-T cells infusion: 30-60 minutes before infusion, H1 anti-histamine agents are applied (acetaminophen 30mg,po.; promethazine 25mg,i.v. ; diphenhydramine 0.5-1mg/kg, no more than 50mg.). Non-physiological doses of corticosteroids are not applied for patients during treatment or recovery unless a life-threatening emergency occurs. CD19 CAR-T cells are infused into patients for one time, the number of infused CD19 CAR-T cells are 0.5-4×10^6/kg.

SUMMARY:
To evaluate the safety and efficacy of targeted CD19 chimeric antigen receptor T cell infusion in the treatment of relapsed or refractory CD19 positive non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CD19 positive, relapsed or refractory diffuse large B cell lymphoma and follicular lymphoma who have no effective treatment (such as autologous or allogeneic stem cell transplantation) and have a survival time of several months or less than 2 years must meet all of the following inclusion criteria, and those who do not meet any of the exclusion criteria can be included:

  1. Non Hodgkin's lymphoma was confirmed by histological examination, and one of the following conditions was met:

     1. Relapsed and refractory CD19 positive diffuse large B-cell lymphoma: at least after the standard second-line drug treatment, the efficacy evaluation did not reach partial remission or above, or reached partial remission or disease progression after partial remission, or relapsed after complete remission;
     2. Relapsed and refractory CD19 positive follicular lymphoma: at least after the standard three-line drug treatment, the efficacy evaluation did not reach partial remission or above, or reached partial remission and disease progress after partial remission, or relapsed after complete remission;
     3. Relapsed refractory CD19 positive diffuse large B-cell lymphoma and follicular lymphoma: primary drug resistance; relapse within 1 year after autologous stem cell transplantation only, not affected by other treatment methods previously used; CD20 positive patients should receive corresponding targeted treatment;
  2. Age: 18-65 years (including boundary value), gender unlimited;
  3. The expected survival time was more than 3 months;
  4. ECOG score 0-1 (dose increasing stage), ECoG score 0-2 (expanding group stage);
  5. The functions of liver and kidney, heart and lung meet the following requirements:

     ① Creatinine ≤ 1.5 ULN

     ②ALT/AST ≤2.5 ULN；

     ③ Total bilirubin ≤ 1.5 × ULN;

     ④ Baseline oxygen saturation ≥ 92%;

     ⑤ No pericardial effusion was detected by echo;
  6. According to Lugano's response standard, there should be at least one measurable tumor focus;
  7. Be able to understand the test and have signed the informed consent.

Exclusion Criteria:

1. Before screening, they received other chimeric antigen receptor therapy or gene modified cell therapy;
2. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) is positive and the DNA titer of peripheral blood hepatitis B virus (HBV) is not within the normal reference range; hepatitis C virus (HCV) antibody is positive and peripheral blood HCV RNA is positive; human immunodeficiency virus (HIV) antibody is positive; cytomegalovirus (CMV) DNA is positive; syphilis is positive ;
3. Subjects who were undergoing systemic steroid therapy at the time of screening and who were determined by the investigator to require long-term systemic steroid therapy during the treatment (except for inhalation or local use);
4. In addition to cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical operation, and breast ductal carcinoma in situ after radical operation, malignant tumors other than B-cell acute lymphoblastic leukemia in the first 5 years were screened;
5. Subjects with graft-versus-host disease (GVHD), autoimmune diseases (such as rheumatoid arthritis, systemic lupus erythematosus and Crohn's disease) and / or requiring immunosuppressant within 2 years;
6. Any unstable heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (NYHA classification ≥ grade III) and severe arrhythmia;
7. Any unstable systemic diseases: including but not limited to liver, kidney or metabolic diseases requiring drug treatment;
8. Subjects who received stem cell transplantation within 6 weeks after CD19 car-t infusion were planned;
9. Invasion of central nervous system;
10. Pregnant women and lactating women; and female subjects who plan pregnancy within 1 year after cell transfusion or male subjects whose partners plan pregnancy within 1 year after cell transfusion;
11. According to the judgment of the researchers, it does not conform to the situation of cell preparation;
12. Other researchers think it's not suitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
BORR | 6 months
  Best objective response rate

SECONDARY OUTCOMES:
Incidence of AE | 2 years
  Incidence of adverse reactions
Pharmacokinetic parameters | 90 Days
  the area under the curve of 28 days AUC0-28d and 90 days AUC0-90d of targeting CD19 chimeric antigen receptor T cells in peripheral blood after administration
Overall survival time | through study completion, an average of 5 year
  Overall survival time
Duration of remission after administration | through study completion, an average of 5 year
  Duration of remission after administration
Disease progression free survival | through study completion, an average of 5 year
  Disease progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided